CLINICAL TRIAL: NCT04718077
Title: Effectiveness of Intraosseous Injection of Dexamethasone Following Impacted Mandibular Third Molar Removal (Randomized Controlled Clinical Trial)
Brief Title: Intraosseous vs Submucosal Injection of Dexamethasone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Corticosteriod
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Tooth, Impacted
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IO dexamethasone injection (Experimental)
  Interventions: Other: Intraosseus
- SM dexamethasone injection. (Active Comparator)
  Interventions: Other: Submucoal

INTERVENTIONS:
Other: Intraosseus — IO dexamethasone injection Dexamethasone 4 mg
  Arms: IO dexamethasone injection
Other: Submucoal — SM dexamethasone injection Dexamethasone 4 mg
  Arms: SM dexamethasone injection.

SUMMARY:
Thirty-eight patients were randomly divided into 2 groups; the intraosseous injection group of dexamethasone (4 mg) and the submucosal injection group. All surgeries were performed by one surgeon.

Postoperative pain was evaluated by visual analog scale score immediately after surgery and on postoperative days 1, 3, and 7.

Swelling (determined using two linear measurements) were assessed just before the surgery and on postoperative days 1, 3, and 7 by using a digital vernier caliper.

Early healing of periodontal soft tissue wound was assessed by using Early Wound Healing Score (EHS) which composed of 3 parameters: clinical signs of re-epithelization (CSR), clinical signs of hemostasis (CSH), and clinical signs of inflammation (CSI) and were assessed on postoperative days 1, 7, and 14. Mouth opening (determined by measurement of the maximum inter-incisal distance) were assessed just before the surgery and on postoperative days 1, 3, and 7 by using a digital vernier caliper.

ELIGIBILITY:
Inclusion criteria

* Patient complaining of impacted mandibular third molar mesioangular or horizontal, according to the Pell and Gregory classification 1933)
* Healthy patient (American society of anesthesiologists class I status)
* Patient age range from 18 to 40 years old.
* Patient without any local inflammation or pathology.
* Patient who will able to understand verbal and written instructions.

Exclusion criteria

* Pregnant or breast-feeding women.
* Patient had anti-inflammatory drugs within 2 weeks before the procedure.
* Patient under radiotherapy or chemotherapy.
* Habits (heavy smoking and alcoholic).
* Allergy to drugs used in this study.
* Patient under anticoagulant or corticosteroid therapy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change in mouth opening | baseline, 1st, 3rd, 7th days
  determined by measurement of the maximum inter-incisal distance assessed by using a digital vernier caliper
change in swelling | 1st, 3rd, 14th days
  assessed by measuring two linear references (horizontal and vertical) with digital vernier caliper
  1. Horizontal reference between the corner of the mouth and the tragus of the ear.
  2. Vertical reference between the lateral canthus and the angle of the mandible.
change in pain scores | 1st, 3rd, 7th days
  Pain will be assessed by using a visual analog scale (VAS) (13) immediately after surgery and on postoperative days 1, 3, and 7.

SECONDARY OUTCOMES:
change in early healing of periodontal soft tissue wound | 1st, 7th, 14th days
  The EHS is composed of 3 parameters:
  1. Clinical signs of re-epithelization (CSR).
  2. Clinical signs of haemostasis (CSH).
  3. Clinical signs of inflammation (CSI).

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Azarita, Egypt